CLINICAL TRIAL: NCT00081887
Title: Phase I Study of Weekly Clofarabine for the Treatment of Relapsed/Refractory Chronic Lymphocytic Leukemia
Brief Title: Study of Weekly Clofarabine for the Treatment of Relapsed/Refractory Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0134
Record Dates: First submitted 2004-04-23; First posted 2004-04-27 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Leukemia; Clofarabine; Clofarex; Clolar
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weekly Clofarabine (Experimental)
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Starting dose is 10 mg/m^2 as a 1-hour infusion into a vein once every 2 weeks for 4 weeks (1 cycle).
  Other Names: Clofarex; Clolar

SUMMARY:
Primary Objectives:

1. To determine the maximum tolerated dose (MTD) of clofarabine in Chronic Lymphocytic Leukemia (CLL).
2. To determine the toxicity profile of clofarabine in CLL.
3. To investigate the plasma clofarabine and cellular clofarabine triphosphate pharmacology profile of clofarabine in CLL.

DETAILED DESCRIPTION:
Clofarabine is a new chemotherapy drug that is designed to interfere with the growth and development of cancer cells.

Before you can start treatment on the study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical examination. You will also be asked about what medications you are taking currently and about the level of your daily activities. Routine blood tests (about 2 tablespoons) will be done within 14 days before the start of the study to make sure that you are not at increased risk for developing side effects. You may have bone marrow samples collected. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle.

If you are found to be eligible, you will receive clofarabine as a 1-hour infusion into a vein once once every 2 weeks for 4 weeks. This cycle makes up one treatment course.

The drug is evaluated at different dose levels. The first three patients will start with a lower dose. Unless serious side effects occur, the next group of patients (usually groups are 3 patients, although they can be expanded to include more patients if needed) will receive a higher dose.

If you show a response and do not experience any severe side effects, you can receive up to a total of 6 courses of therapy. During each course, clofarabine is given the same way as during the first course. However, the dose of clofarabine may be lowered during later courses to decrease the risk of side effects that may have occurred in previous courses. If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

Before every treatment course, your doctor will perform a physical exam, including measurement of your weight and vital signs. You will be asked about the level of your daily activities and how you are feeling. At least once every two weeks (more often if your doctor feels it is necessary), you will have blood samples (about 1-2 teaspoons) collected for routine lab tests. Repeat bone marrows will be collected after the third and sixth course. However, if you complete the study before the third course, the bone marrow may be taken then. No bone marrow may be taken if the condition of your disease is obvious from the blood.

You will need to stay in Houston for the first 4 weeks of treatment. After that, you may return to your home but you will still have to return to Houston to receive the clofarabine treatment. You may choose to have check-up visits and blood tests with your local doctor.

After you finished your treatment, and as long you are participating on this study, you will be scheduled every 3-6 months to check on the status of the disease and your overall health.

This is an investigational study. Clofarabine is authorized by the FDA for use in research only. Up to 36 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic lymphocytic leukemia (CLL), CLL/PLL (as defined by FAB), and PLL (B- and T-cell phenotypes) who have relapsed from or are refractory to at least one fludarabine-based regimen.
2. Absolute neutrophil count (ANC) >= 1 x 10(9)/L and platelet count >= 50 x 10(9)/L
3. Adequate liver function (total bilirubin <= 1.5 x ULN, SGPT <= 2.5 x ULN) and renal function (serum creatine <= 1.5 x ULN).
4. ECOG performance status <= 2.

Exclusion Criteria:

1. Patients with NYHA >= grade 3 heart disease as assessed by history and/or physical examination
2. Pregnant or breastfeeding women or patients who are unwilling or unable to practice adequate contraception.
3. Chemotherapy within 4 weeks of starting therapy, or concurrent anticancer therapy (chemotherapy, radiotherapy, or biologic therapy)
4. Other malignancy within 3 years except in situ carcinoma
5. Unwilling or unable to provide informed consent
6. Hypersensitivity to nucleoside analogues
7. Other significant medical condition that compromises safety, compliance or study conduct, including but not limited to uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within 6 months, ventricular arrhythmia, diabetes, active infection, pulmonary fibrosis, and chronic hepatitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-05; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Following each 4 week treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Faderl, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org